CLINICAL TRIAL: NCT03660657
Title: Effectiveness and Cost-effectiveness of Ozone Therapy in Patients With Ischemic Heart Disease Refractory to Medical and Surgical Treatment: Randomized, Triple-blind Clinical Trial
Brief Title: Ozone Therapy in Refractory Ischemic Heart Disease.
Acronym: O3Cardio
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Very low recruitment. During COVID-19 pandemic these are patients of high risk.
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Servicio Canario de Salud (Other); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Fundación Canaria de Investigación Sanitaria (Other); Colegio Oficial de Médicos de Las Palmas (Unknown); Fundación MAPFRE Guanarteme (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, MD, PhD, Head of Research Unit, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: O3Cardio; 2018-000201-24 (EudraCT Number); 2018-000201-24 (Other: Registro Español de Ensayos Clínicos (REec)); PIFUN44/17 (Other Grant/Funding Number: Fundación Canaria de Investigación Sanitaria (FUNCANIS))
Record Dates: First submitted 2018-08-23; First posted 2018-09-06 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Heart Disease
Keywords: complementary and integrative medicine; cost-effectiveness ratio; ischemic heart disease; heart failure; ozone therapy; quality of life related to health; shared decision-making tool
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure | interventions — Ozone; Oxygen

STUDY DESIGN:
Intervention Model Description: Standard treatment + ozone therapy (O3/O2) versus Standard treatment + oxygen (O2) as placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of: patients, cardiologist and cardiac surgeons (clinical assessment), investigators obtaining other parameters (quality of life, biochemical and clinical parameters), investigators for statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone Group: (Experimental): Standard treatment + Ozone therapy (O3/O2)
  Interventions: Drug: Ozone
- Control Group: (Placebo Comparator): Standard treatment + Oxygen (O2)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Ozone — Ozone Group: Standard treatment + Ozone therapy (O3/O2) by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 µg/ml; 40 sessions in 16 weeks.
  Other Names: O3
  Arms: Ozone Group:
Drug: Oxygen — Control Group: Standard treatment + Oxygen (O2) by rectal insufflation. O3/O2 concentration = 0 µg/ml (only O2); 40 sessions in 16 weeks.
  Other Names: O2
  Arms: Control Group:

SUMMARY:
The main objective of this clinical trial is to evaluate the effectiveness and cost-effectiveness of adding ozone therapy to standard management of patients with advanced ischemic heart disease refractory to medical and surgical treatment.

DETAILED DESCRIPTION:
This study will evaluate the potential role of ozone therapy added to the standard management of patients with symptomatic refractory ischemic heart disease, III-IV functional class of the classification of the New York Heart Association (NYHA).

MAIN OBJECTIVES: 1) to evaluate clinical effect and quality of life related to health (HRQOL) of adding O3 to the standard treatment of these patients. 2) to estimate the additional costs of adding O3 to the standard treatment and to evaluate the cost-effectiveness ratio.

SECONDARY OBJECTIVES: 3) To evaluate the evolution of a) biochemical parameters; b) cardiovascular parameters; c) toxicity of O3. 4) Develop and evaluate the acceptability of a shared decision-making (SDM) tool between professionals and patients.

METHODOLOGY: Phase II-III clinical trial, randomized, triple-blind. Sample size: 18 patients.

TREATMENT: All patients will receive their standard treatment + 40 sessions of rectal insufflation:

1. Ozone-Group (n = 9): O3/O2 concentration progressively increased from 10 to 30 µg/ml.
2. Control-placebo-Group (n = 9): O3/O2 Concentration = 0 µg/ml (only O2).

Main Variables: 1) changes in the self-perceived quality of life (Minnesota scale). 2) Direct costs.

Secondary Variables: 1) biochemical parameters; 2) Cardiovascular parameters; 3) Side effects. 4) acceptability of patients to a shared decision-making (SDM) tool.

Length of treatment: 16 weeks.

Follow-up: 16 weeks after completion of O3.

Assessments: 1) Pre-O3 (basal), 2) pos-O3 (end of O3), 3) 4 months pos-O3.

Planned length of clinical trial: 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ischemic heart disease, Functional Class III-IV from the NYHA, with symptoms in spite of maximal conventional medical treatment and no suitable to further percutaneous or surgical procedures.
* It should be required clinical diagnosis by the Cardiology Department and confirmation by cardiac catheterization with coronary angiography.
* Ejection Fraction < 40%
* Patients who have signed and dated the study 's specific informed consent.
* Before enrollment, women of childbearing potential should obtain a negative result in the serum or urine pregnancy test at the screening visit, and accept the use of appropriate contraceptive methods at least from the 14 days prior to the first dose of the study drug. up to 14 days after the last one.

Exclusion Criteria:

* Age < 18 or > 85 years old.
* Severe valve disease and/or dynamic left ventricular outflow tract obstruction.
* Pregnancy at the time of enrollment.
* Limited walking ability due to neurologic or orthopedic impairments of the legs
* Those who are incapable to fill in the scales used to measure the quality of life variables
* Cerebral vascular accident (CVA or Transient Ischemic Attack (TIA) within the previous 3 months or carotid stenosis > 80%.
* Acute myocardial infarction (AMI), Percutaneous coronary intervention (PCI) or transmyocardial laser revascularization (TMR or PMR) within the previous 3 months.
* Hemodynamically or clinically unstable patients.
* Severe or limiting pulmonary diseases.
* Specific liver enzymes [Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) > 5 times the upper limit of normal
* Increased creatinine > 3 times the upper limit of normal or Glomerular Filtration Rate (GFR) < 25 ml/min or who are on chronic renal dialysis.
* Severe peripheral vascular disease with rest pain or significant chronic wounds.

Uncontrolled cancer disease or severe active systemic infection or HIV.

* Life expectancy < 4 months
* Contraindication or disability for rectal ozone administration or to attend scheduled treatments.
* Known allergy to ozone.
* Patients who do not meet all the inclusion criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of 21 physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. Each item is scored from 0 (no affected) to 5 (very much affected). Total range from 0 (best) to 105 (worst)
Direct Hospital Cost (at the end of ozone therapy) | 16 weeks
  The direct expenses incurred by the hospital in providing services (medication, tests, medical visits...) during the 16 weeks of ozone therapy (in euros).

SECONDARY OUTCOMES:
Change from Baseline in quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in quality of life by the "Short Form 36-item health survey" (SF-36) questionnaire (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of 36 items (0 = worst, 100 = best). Final accumulated total range from 0 (worst) to 100 (best)
Change from Baseline in Montreal Cognitive Assessment (MOCA) questionnaire (at the end of ozone therapy) | 16 weeks
  Assessment of 8 types of cognitive abilities by a total 30-point test (0 = worst, 30 = best)
Change from Baseline in Biochemical cardiac parameters (High sensitive troponin, pro-brain natriuretic peptide (proBNP)) (at the end of ozone therapy) | 16 weeks
  Serum levels of high sensitive troponin and proBNP
Change from Baseline in Biochemical parameters of oxidative stress (at the end of ozone therapy) | 16 weeks
  Serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals
Change from Baseline in Biochemical parameters of inflammation (at the end of ozone therapy) | 16 weeks
  Serum levels of pro-inflammatory interleukins and TNFalpha
Change from Baseline (by Echocardiograpy) of: left ventricular end-diastolic volume (LVEDV) and left ventricular end-systolic volume (LVESV) (at the end of ozone therapy) | 16 weeks
  Measurement of volume (in ml) of LVEDV and LVESV.
Change from Baseline (by Echocardiograpy) of left ventricular ejection fraction (LVEF) (at the end of ozone therapy) | 16 weeks
  Measurement (in percentage) of LVEF
Change from Baseline in Six-minute walk test (6MWT) (at the end of ozone therapy) | 16 weeks
  Assessment of functional exercise capacity according to the walking distance covered over a time of 6 minutes (in meters)
Change from Baseline in cerebral blood flow by Transcranial doppler (at the end of ozone therapy) | 16 weeks
  Doppler ultrasound evaluation of systolic and diastolic velocity in middle cerebral arteries (in cm/s)
Change from Baseline in Hyperspectral image of the supraciliary area (at the end of ozone therapy) | 16 weeks
  Assessment of the percentage of reflectance for each wavelength
Change from Baseline in lower limb blood flow by Doppler ultrasound (at the end of ozone therapy) | 16 weeks
  Doppler ultrasound evaluation of systolic and diastolic velocity in lower limbs (in cm/s)
Change from Baseline in Hyperspectral image of lower limbs (at the end of ozone therapy) | 16 weeks
  Assessment of the percentage of reflectance for each wavelength
Incidence of severe adverse events in accordance with the definition of the Council for International Organizations of Medical Sciences (at the end of ozone therapy) | 16 weeks
  Number of events that are fatal, life threatening, leading to or prolonging a stay in hospital, or resulting in severe disability
Quality of Life (QoL) measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) (at 32 weeks) | 32 weeks
  Self-reported evaluation of 21 physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. Each item is scored from 0 (no affected) to 5 (very much affected). Total range from 0 (best) to 105 (worst)
Direct Hospital Cost (at 32 weeks) | 32 weeks
  The direct expenses incurred by the hospital in providing services (medication, tests, medical visits...) during the 16 weeks of ozone therapy (in euros)
Change from Baseline in quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire (at 32 weeks) | 32 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in quality of life by the "Short Form 36-item health survey" (SF-36) questionnaire (at 32 weeks) | 32 weeks
  Self-reported evaluation of 36 items (0 = worst, 100 = best). Final accumulated total range from 0 (worst) to 100 (best)
Change from Baseline in Montreal Cognitive Assessment (MOCA) questionnaire (at 32 weeks) | 32 weeks
  Assessment of 8 types of cognitive abilities by a total 30-point test (0 = worst, 30 = best)
Change from Baseline in Biochemical cardiac parameters (High sensitive troponin, pro-brain natriuretic peptide (proBNP)) (at 32 weeks) | 32 weeks
  Serum levels of high sensitive troponin and proBNP
Change from Baseline in Biochemical parameters of oxidative stress (at 32 weeks) | 32 weeks
  Serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals
Change from Baseline in Biochemical parameters of inflammation (at 32 weeks) | 32 weeks
  Serum levels of pro-inflammatory interleukins and TNFalpha
Change from Baseline (by Echocardiograpy) of: left ventricular end-diastolic volume (LVEDV) and left ventricular end-systolic volume (LVESV) (at 32 weeks) | 32 weeks
  Measurement of volume (in ml) of LVEDV and LVESV.
Change from Baseline (by Echocardiograpy) of left ventricular ejection fraction (LVEF) (at 32 weeks) | 32 weeks
  Measurement (in percentage) of LVEF
Change from Baseline in Six-minute walk test (6MWT) (at 32 weeks) | 32 weeks
  Assessment of functional exercise capacity according to the walking distance covered over a time of 6 minutes (in meters)
Change from Baseline in cerebral blood flow by Transcranial doppler (at 32 weeks) | 32 weeks
  Doppler ultrasound evaluation of systolic and diastolic velocity in middle cerebral arteries (in cm/s)
Change from Baseline in Hyperspectral image of the supraciliary area (at 32 weeks) | 32 weeks
  Assessment of the percentage of reflectance for each wavelength
Change from Baseline in lower limb blood flow by Doppler ultrasound (at 32 weeks) | 32 weeks
  Doppler ultrasound evaluation of systolic and diastolic velocity in lower limbs (in cm/s)
Change from Baseline in Hyperspectral image of lower limbs (at 32 weeks) | 32 weeks
  Assessment of the percentage of reflectance for each wavelength
Incidence of severe adverse events in accordance with the definition of the Council for International Organizations of Medical Sciences (at 32 weeks) | 32 weeks
  Number of events that are fatal, life threatening, leading to or prolonging a stay in hospital, or resulting in severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Dr. Negrín University Hospital, Las Palmas, Spain; Pedro G Serrano-Aguilar, MD, PhD, Study Director — Servicio de Evaluación. Servicio Canario de Salud. Spain; Renata Linertová, PhD, Principal Investigator — Servicio de Evaluación. Servicio Canario de Salud. Spain; Bernardino Clavo, MD, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Celestina Amador, MD, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Francisco Rodríguez-Esparragón, BSc, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Norberto Santana-Rodríguez, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center, Riyadh, Kingdom of Saudi Arabia
Locations (1):
- Dr. Negrin University Hospital, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buyuklu M, Kandemir FM, Set T, Bakirci EM, Degirmenci H, Hamur H, Topal E, Kucukler S, Turkmen K. Beneficial Effects of Ozone Therapy on Oxidative Stress, Cardiac Functions and Clinical Findings in Patients with Heart Failure Reduced Ejection Fraction. Cardiovasc Toxicol. 2017 Oct;17(4):426-433. doi: 10.1007/s12012-017-9400-8. PMID 28097518
- [Background] Bocci V, Borrelli E, Travagli V, Zanardi I. The ozone paradox: ozone is a strong oxidant as well as a medical drug. Med Res Rev. 2009 Jul;29(4):646-82. doi: 10.1002/med.20150. PMID 19260079
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Clavo B, Perez JL, Lopez L, Suarez G, Lloret M, Rodriguez V, Macias D, Santana M, Morera J, Fiuza D, Robaina F, Gunderoth M. Effect of ozone therapy on muscle oxygenation. J Altern Complement Med. 2003 Apr;9(2):251-6. doi: 10.1089/10755530360623365. PMID 12804078
- [Background] Clavo B, Catala L, Perez JL, Rodriguez V, Robaina F. Ozone Therapy on Cerebral Blood Flow: A Preliminary Report. Evid Based Complement Alternat Med. 2004 Dec;1(3):315-319. doi: 10.1093/ecam/neh039. Epub 2004 Oct 6. PMID 15841265
- [Background] Clavo B, Eltobgy K, Caballero E, Abad C, Rodriguez-Esparragon F, Santana-Rodriguez N. Is There a Place for Ozone Therapy in Patients with Heart Failure? Cardiovasc Toxicol. 2017 Oct;17(4):496-497. doi: 10.1007/s12012-017-9423-1. No abstract available. PMID 28853025
- [Background] Di Filippo C, Marfella R, Capodanno P, Ferraraccio F, Coppola L, Luongo M, Mascolo L, Luongo C, Capuano A, Rossi F, D'Amico M. Acute oxygen-ozone administration to rats protects the heart from ischemia reperfusion infarct. Inflamm Res. 2008 Oct;57(10):445-9. doi: 10.1007/s00011-008-7237-0. PMID 18827966
- [Background] Giunta R, Coppola A, Luongo C, Sammartino A, Guastafierro S, Grassia A, Giunta L, Mascolo L, Tirelli A, Coppola L. Ozonized autohemotransfusion improves hemorheological parameters and oxygen delivery to tissues in patients with peripheral occlusive arterial disease. Ann Hematol. 2001 Dec;80(12):745-8. doi: 10.1007/s002770100377. Epub 2001 Oct 13. PMID 11797116
- [Background] Martinez-Sanchez G, Delgado-Roche L, Diaz-Batista A, Perez-Davison G, Re L. Effects of ozone therapy on haemostatic and oxidative stress index in coronary artery disease. Eur J Pharmacol. 2012 Sep 15;691(1-3):156-62. doi: 10.1016/j.ejphar.2012.07.010. Epub 2012 Jul 13. PMID 22796450
- [Background] Bocci V, Zanardi I, Travagli V. Ozone: a new therapeutic agent in vascular diseases. Am J Cardiovasc Drugs. 2011;11(2):73-82. doi: 10.2165/11539890-000000000-00000. PMID 21446774
- See also: EU Clinical Trials Register (European Union Clinical Trials Register) — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2018-000201-24
- See also: Spanish Clinical Studies Registry — https://reec.aemps.es/reec/public/list.html